CLINICAL TRIAL: NCT01287416
Title: Circle of Life.Improving Capacity of Swampy Cree Community Members to Recognize People at Risk for Suicide: A Randomized Controlled Pilot Study
Brief Title: Circle of Life. Improving Capacity of Swampy Cree Community Members to Recognize People at Risk for Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Jitinder Sareen, Professor, Department of Psychiatry, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H2010:192
Record Dates: First submitted 2011-01-10; First posted 2011-02-01 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Suicide
Keywords: Suicide Intervention; Applied Suicide Intervention Skills Training (ASIST); Resilience Retreat; First Nations; Suicide Intervention and Response Inventory (SIRI)
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Applied Suicide Intervention Skills Training (ASIST) (Experimental): ASIST is a 2-day intensive, interactive and practice-dominated course aimed at enabling people to recognize risk and learn how to intervene immediately to prevent suicide. The training is designed for anyone (especially those in a position of trust), from professionals and volunteers to members of the community. Participants range from those in caring roles to people concerned about family members or friends. The theory is that suicide can be pre¬vented with the help of prepared caregivers. ASIST is designed to help all caregivers become more willing, ready and able to help persons at risk. Just as "CPR" skills make physical first aid possible, training in suicide intervention develops the skills used in suicide first aid.
  Interventions: Behavioral: Applied Suicide Intervention Skills Training
- Resilience Retreat (Active Comparator): The two days will be divided into cultural activities, sharing circles, small group discussions, story telling and dance. Two First Nations community leaders will be identified to lead each of the two retreats.
  Interventions: Behavioral: Resilience Retreat

INTERVENTIONS:
Behavioral: Applied Suicide Intervention Skills Training — Applied Suicide Intervention Skills Training (ASIST) is a 2-day, 14 hour suicide intervention skills training workshop.
  Other Names: ASIST
  Arms: Applied Suicide Intervention Skills Training (ASIST)
Behavioral: Resilience Retreat — The Resilience Retreat is a 2-day, 14 hour session
  Arms: Resilience Retreat

SUMMARY:
Primary Hypothesis: Participants in the Applied Suicide Intervention Skills Training (ASIST) gatekeeper training will be significantly more likely to have increased knowledge and preparedness to help people with suicidal ideation than participants who receive the resilience retreat.

Secondary Hypotheses:

1. Participants in ASIST gatekeeper training will not have higher levels of post-intervention distress or suicidal ideation compared to the resilience retreat.
2. High levels of distress, grief, and alcohol abuse will significantly impact on the learning and retention of suicide intervention skills.

DETAILED DESCRIPTION:
Inclusion criterion: All members of the Swampy Cree Tribal communities who are currently residing on the reserves will be eligible to participate in the study.

Exclusion criterion: Exclusion criteria for the study include being less than 16 years of age, prior training in SafeTALK or ASIST, being an elected official in a First Nations community, and inability to read or write.

Primary outcome: Skills in Suicide Intervention: Suicide Intervention Response Inventory.The Suicide Intervention Response Inventory (SIRI) will be used to detect enhancement of intervention skills in participants. The SIRI is a self-administered test that was designed to measure competence in choosing appropriate response to a series of clinical scenarios with suicidal individuals. Research on the SIRI has shown its good psychometric properties, freedom from social desirability effects, and responsiveness to training in suicide prevention. It contains 25 items, each of which consists of a "client" remark and two "helper" responses. Responses are judged based on response options made by highly expert suicidologists. The SIRI has shown good internal consistency with alpha of 0.834, and good test-retest reliability.

Secondary Outcomes:

* Knowledge about suicide, attitudes toward suicide, and self-reported preparedness to intervene with suicidal behavior will be measured by a series of questions that were developed by LivingWorks Inc.
* Gatekeeper behaviors will be measured similar to questions utilized by Wyman in the school-based study that assess how many people had the person asked others about suicide.

ELIGIBILITY:
Inclusion Criteria:

* All members of the Swampy Cree Tribal communities who are currently residing on the reserves will be eligible to participate in the study.

Exclusion Criteria:

* being less than 16 years of age
* prior training in SafeTALK or ASIST
* being an elected official in a First Nations community

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jitender Sareen, MD, Principal Investigator — Department of Psychiatry, Faculty of Medicine, University of Manitoba
Locations (1):
- University of Manitoba Department of Psychiatry, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Sareen J, Isaak C, Bolton SL, Enns MW, Elias B, Deane F, Munro G, Stein MB, Chateau D, Gould M, Katz LY. Gatekeeper training for suicide prevention in First Nations community members: a randomized controlled trial. Depress Anxiety. 2013 Oct;30(10):1021-9. doi: 10.1002/da.22141. Epub 2013 Jun 12. PMID 23761133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Various methods of advertising for volunteers was used (i.e., radio advertisements, newsletters, posters). Community activities were organized by community representatives in an effort to recruit individuals to participate in the study (i.e., through a bingo night, barbecue, etc.) between May 2010 and May 2011.
Pre-assignment Details: From all eligible applications, we selected participants using a random number generator based on receipt of application until we had six adolescents, four adults, and two elders in each community who met criteria for participation in the study.
Groups:
- Applied Suicide Intervention Skills Training (ASIST): Applied Suicide Intervention Skills Training (ASIST) is a 2-day, 14 hour suicide intervention skills training workshop. ASIST is an intensive, interactive and practice-dominated course aimed at enabling people to recognize risk and learn how to intervene immediately to prevent suicide. The training is designed for anyone (especially those in a position of trust), from professionals and volunteers to members of the community. Participants range from those in caring roles to people concerned about family members or friends. The theory is that suicide can be pre¬vented with the help of prepared caregivers. ASIST is designed to help all caregivers become more willing, ready and able to help persons at risk. Just as "CPR" skills make physical first aid possible, training in suicide intervention develops the skills used in suicide first aid.
- Resilience Retreat: The 2-day 14-hour resilience retreat (RR) was divided into cultural teachings and activities, sharing circles, small group discussions, and story telling. The RR included four main components: (1) Seven Sacred Teachings; (2) Self-identity-focused on knowing your identity, the past, and celebrating your history. Following the presentation, participants divided into community groups for discussion and then reconvened with all attendees to share discussion points; (3) Healthy communities-explored and discussed questions regarding healthy communities using both verbal and pictorial explanations; (4) Bracelet-making activity. The RR ended with a sharing circle attended by all participants.
Period: Pre-post Training
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Started | 48 (number of people that were invited to participate based on eligibility and consent received) | 48 (number of people that were invited to participate based on eligibility and consent received)
Training Workshop | 31 (number of people that showed up for the training session) | 24 (number of people that showed up for the training session)
Post Training Questionnaire | 26 | 23
Completed | 26 | 23
Not Completed | 22 | 25
Not completed — Withdrawal by Subject | 17 | 24
Not completed — Lost to Follow-up | 5 | 1
Period: 6 Month Follow-up
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Started | 31 (all participants that had completed the baseline measure were invited to do the follow-up) | 24 (all participants that had completed the baseline measure were invited to do the follow-up)
Completed | 28 | 22
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: The number of baseline participants reflects the number of participants that showed up on the day of training, as that was our first point of contact and the time point at which the baseline questionnaire was given. This is different than the number of people that we invited to participate in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat | Total
Number analyzed (Participants) | 31 | 24 | 55
Age, Customized [Number; unit: participants]
  16-21 | 15 | 9 | 24
  22-44 | 8 | 10 | 18
  45+ | 8 | 4 | 12
  Missing | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 33
  Male | 10 | 12 | 22
Marital status [Number; unit: participants]
  Never married | 12 | 14 | 26
  Widowed/separated/divorced | 4 | 3 | 7
  Married/common-law | 11 | 7 | 18
  Missing | 4 | 0 | 4
Educational attainment [Number; unit: participants] — Level of educational attainment of the participant
  participants
    Grade 9 or lower | 19 | 3 | 22
    Grade 10 or higher | 12 | 21 | 33
Language spoken most often [Number; unit: participants]
  English | 20 | 20 | 40
  Cree | 9 | 4 | 13
  Missing | 2 | 0 | 2
Current work status [Number; unit: participants]
  Working full- or part-time | 6 | 8 | 14
  Unemployed/social assistance | 14 | 11 | 25
  Retired/at home full-time/student | 11 | 5 | 16
Know someone who died by suicide [Number; unit: participants]
  Yes | 28 | 21 | 49
  No | 3 | 3 | 6
When most recent suicide death [Number; unit: participants] — measured only among those who had reported knowing someone who died by suicide
  participants
    More than 1 year ago | 18 | 10 | 28
    Within the last year | 3 | 8 | 11
    Within the last 6 months | 5 | 3 | 8
    Within the last 1 month | 0 | 0 | 0
    Missing | 2 | 0 | 2
    Did not know someone who died by suicide | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: SIRI Questionnaire Score
Description: The Suicide Intervention Response Inventory (SIRI-2) will be used to detect enhancement of intervention skills in participants. The 25-item SIRI-2 is a self-administered test that was designed to measure competnce in choosing appropriate response to a series of clinical scenarios with suicidal individuals. Research on the SIRI-2 has shown its good psychometric properties, freedom from social desirabiity effects and responsiveness to training in suicide prevention.
Time Frame: pre-training, post-training and 6 mo follow up
Measure: Mean (Standard Deviation); unit: number of items correct
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
number of items correct
  Pre-training | 12.90 (2.78) | 14.17 (4.10)
  Post-training | 14.83 (3.92) | 14.30 (3.42)
  6 month follow-up | 13.52 (3.72) | 15.05 (3.58)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; The null hypothesis was that the groups would not differ in terms of SIRI scores across the three time points. We used linear mixed models to determine whether scores were different between the two groups over time; Test type: Superiority or Other; p = 0.61, Mixed Models Analysis — The a priori threshold for statistical significance was set at p<.05. Effect size determined by partial eta-squared to be 0.01; Model was adjusted for differences in educational attainment at baseline

2. Secondary Outcome: Self-perceived Confidence in Helping a Suicidal Individual
Description: Meaures the level of confidence that the individual believes they have in helping a suicidal person based on a 4 point Likert scale ranging from 1 (not at all confident) to 4 (very confident).
Time Frame: pre-training, post-training and 6 month follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
scores on a scale
  Pre-training | 2.68 (0.91) | 2.87 (0.80)
  Post-training | 2.73 (0.78) | 2.57 (0.99)
  6 month follow-up | 2.63 (0.93) | 2.68 (0.84)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; The null hypothesis was that the groups would not differ in terms of level of knowledge across the three time points; Test type: Superiority or Other; p = 0.95, Mixed Models Analysis — The a priori threshold for statistical significance was set at p<.05. Effect size determined by partial eta-squared to be 0.02; Model was adjusted for differences in educational attainment at baseline

3. Secondary Outcome: Self-perceived Skill in Helping a Suicidal Individual
Description: Measures the level of ability that the individual believes they have in helping a suicidal person based on a 4 point Likert scale ranging from 1 (not at all skilled) to 4 (very skilled).
Time Frame: pre-training, post-training and 6 month follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
scores on a scale
  Pre-training | 1.94 (0.77) | 2.00 (0.74)
  Post-training | 2.50 (0.76) | 2.23 (0.97)
  6 month follow-up | 2.43 (0.92) | 2.27 (0.97)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; The null hypothesis was that the two groups would not differ in terms of self-reported skill level across the three time points; Test type: Superiority or Other; p = 0.33, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model was adjusted for differences in educational attainment at baseline

4. Secondary Outcome: Self-perceived Knowledge About Suicide
Description: Measures the level of knowledge about suicide that the individual believes they have based on a 4 point Likert scale ranging from 1 (not at all knowledgeable) to 4 (very knowledgeable).
Time Frame: pre-training, post-training and 6 month follow-up
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
Scores on a scale
  Pre-training | 2.16 (0.97) | 2.09 (0.79)
  Post-training | 2.65 (0.75) | 2.23 (0.92)
  6 month follow-up | 2.50 (0.88) | 2.23 (0.81)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; The null hypothesis was that the groups would not differ in terms of level of knowledge across the three time points; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — The a priori threshold for statistical significance was set at p<.05. Effect size determined by partial eta-squared to be 0.05; Model adjusted for differences in educational attainment at baseline

5. Secondary Outcome: Self-perceived Preparedness
Description: Measures the level of preparedness of the individual to help someone who is suicidal based on a 4 point Likert scale ranging from 1 (not at all prepared) to 4 (very prepared).
Time Frame: pre-training, post-training and 6 month follow-up
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
Scores on a scale
  Pre-training | 2.19 (0.87) | 2.33 (0.76)
  Post-training | 2.77 (0.91) | 2.39 (0.84)
  6 month follow-up | 2.43 (0.96) | 2.45 (0.86)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; The null hypothesis was that the two groups would not differ on level of self-reported preparedness to help a suicidal person; Test type: Superiority or Other; p = 0.63, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Model was adjusted for differences in educational attainment at baseline

6. Secondary Outcome: Self-reported Distress
Description: Measures the level of distress in the participant using the K6 distress scale. The scale is comprised of six questions which are scored from 0 (none of the time) to 4 (all of the time). The sum of the scores from all six questions was used to determine a total scale score which ranges from 0 (not at all distressed) to 24 (very distressed).
Time Frame: pre-training and 6 month follow-up
Population: The smaller number of participants per group reflects the number of individuals who responded to the baseline and 6 month follow up time point questionnaires.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 28 | 22
Scores on a scale
  Pre-training | 7.62 (0.98) | 6.30 (1.13)
  6 month follow-up | 6.40 (0.80) | 6.77 (0.92)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; The null hypothesis was that the groups would not differ on their level of distress across the two time points; Test type: Superiority or Other; p = 0.21, ANCOVA — A priori threshold for significance set to p<.05; Model adjusted for differences in educational attainment at baseline

7. Secondary Outcome: Self-reported Alcohol Use
Description: Details participants' level of alcohol consumption and if it may be harmful according to the AUDIT. The AUDIT scale is comprised of ten questions with most questions being scored from 0 (never) to 4 (4 or more times per week). The sum of the scores from all ten questions was used to determine a total scale score which ranges from 0 (no risk related to alcohol) to 40 (high risk related to alcohol). Total scores of 8 or more are recommended as indicators of hazardous and harmful alcohol use, as well as possible alcohol dependence.
Time Frame: pre-training and 6 month follow-up
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 28 | 22
Scores on a scale
  Pre-training | 12.14 (2.76) | 9.70 (2.35)
  6 month follow-up | 8.38 (1.86) | 8.76 (1.58)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Null hypothesis was that the groups would not differ in terms of alcohol use across the two time points; Test type: Superiority or Other; p = 0.46, ANCOVA — A priori threshold for significance set at p<.05; Model was adjusted for differences in educational attainment at baseline

8. Secondary Outcome: Self-reported Resiliency Score
Description: Assesses resiliency in the participant according to the Connor-Davidson Resilience Scale, 10-item. The CD-RISC 10 is comprised of ten questions scored from 0 (Not at all true) to 4 (True nearly all of the time). The sum of the scores from all ten questions was used to determine a total scale score which ranges from 0 (low resiliency) to 40 (highly resilient).
Time Frame: pre-training and 6 month follow-up
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 28 | 22
Scores on scale
  Pre-training | 21.78 (1.38) | 28.71 (1.49)
  6 month follow-up | 23.68 (1.21) | 27.82 (1.31)
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; The null hypothesis was that the two groups would not differ in resiliency scores across the follow-up period; Test type: Superiority or Other; p = 0.28, ANCOVA — The a priori threshold for statistical significance was set at p<.05; Model is adjusted for differences in educational attainment at baseline

9. Secondary Outcome: Lifetime Suicidal Ideation at Baseline
Description: Number of people who endorsed having thought about suicide in their lifetime as measured at baseline
Time Frame: July 19-20, 2010
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
participants | 14 | 14
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Test type: Superiority or Other; p = 0.33, Chi-squared — A priori threshold for significance set at p<.05

10. Secondary Outcome: Lifetime Suicide Attempt at Baseline
Description: Number of people who endorsed having made a suicide attempt in their lifetime as measured at baseline
Time Frame: July 19-20, 2010
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
participants | 6 | 6
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Test type: Superiority or Other; p = 0.62, Chi-squared — A priori threshold for significance set at p<.05

11. Secondary Outcome: Suicidal Ideation in Past 2 Days at Baseline
Description: Number of people who endorsed having thought about suicide in the past 2 days as measured at baseline (not at all vs a little to a lot)
Time Frame: July 19-20, 2010
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 31 | 24
participants
  Not at all | 29 | 22
  A little to a lot | 2 | 2
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Test type: Superiority or Other; p = 1.00, Fisher Exact — A priori threshold for significance set to p<.05

12. Secondary Outcome: Number of People With Suicidal Ideation in Past 2 Days Immediately Post Training
Description: Number of people who endorsed having thought about suicide in the past 2 days as measured immediately post training (not at all vs a little to a lot)
Time Frame: July 22-23, 2010
Population: The smaller number of participants per group reflects the number of individuals who responded to the post-training questionnaire.
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 25 | 23
participants
  Not at all | 23 | 21
  A little to a lot | 2 | 2
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Test type: Superiority or Other; p = 1.00, Fisher Exact — A priori threshold for significance set to p<.05

13. Secondary Outcome: Suicidal Ideation Since Training at 6 mo Follow-up
Description: Number of people who endorsed having thought about suicide since the training as measured at 6 month follow-up (not at all vs a little to a lot)
Time Frame: January 28-31, 2011
Population: The smaller number of participants per group reflects the number of individuals who responded to the 6 month follow up time point questionnaire.
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 28 | 22
participants
  Not at all | 21 | 21
  A little to a lot | 7 | 1
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Test type: Superiority or Other; p = 0.064, Fisher Exact — A priori threshold for significance set to p<.05

14. Secondary Outcome: Attempted Suicide Since Training at 6 mo Follow-up
Description: Number of people who endorsed having made a suicide attempt since the training as measured at 6 month follow-up
Time Frame: January 28-31, 2011
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 28 | 22
participants | 0 | 0

15. Secondary Outcome: Gatekeeper Behaviors - Asked Person at Risk About Suicidal Thoughts
Description: Number of participants who have asked someone that they thought was at risk about suicidal thoughts since the training, measured at 6 month follow-up assessment.
Time Frame: January 28-31, 2011
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 28 | 22
participants | 3 | 6
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Null hypothesis was that the groups would not differ in terms of their gatekeeper behaviours; Test type: Superiority or Other; p = 0.14, Fisher Exact — a priori threshold for significance set a p<.05; unadjusted model

16. Secondary Outcome: Gatekeeper Behaviours - Did Not Ask Person at Risk
Description: Number of participants who did not ask someone about their suicidal thoughts even though they thought they were at risk, measured at 6 month follow-up assessment based on time since training.
Time Frame: January 28-31, 2011
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Number analyzed (Participants) | 28 | 22
participants | 9 | 9
Statistical Analysis 1: Comparison: Applied Suicide Intervention Skills Training (ASIST) vs Resilience Retreat; Null hypothesis was that the groups would not differ on gatekeeper behaviours; Test type: Superiority or Other; p = 0.41, Chi-squared — A priori threshold for significance set at p<.05; Unadjusted model

ADVERSE EVENTS:
Time Frame: From baseline time point to 6 months.
Arm/Group | Applied Suicide Intervention Skills Training (ASIST) | Resilience Retreat
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/24
Other Adverse Events (participants affected / at risk) | 0/31 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes